CLINICAL TRIAL: NCT01257594
Title: Pilot Study of EGFR Inhibition Using High Dose Administration of Erlotinib Weekly for Recurrent Malignant Gliomas With EGFR Variant III Mutation
Brief Title: EGFR Inhibition Using Weekly Erlotinib for Recurrent Malignant Gliomas
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Andrew B Lassman, MD (Other)
Collaborators: Genentech, Inc. (Industry); OSI Pharmaceuticals (Industry)
Responsible Party: Sponsor-Investigator, Andrew B Lassman, MD, Associate Professor of Neurology, Columbia University
Organization: Columbia University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AAAJ7500
Record Dates: First submitted 2010-12-08; First posted 2010-12-09 (Estimated); Last update posted 2023-05-25 (Actual); Status verified 2023-05

CONDITIONS: Brain Cancer
Keywords: Gliomas; Erlotinib; Glioblastoma; GBM; Gliosarcoma; Glioma
MeSH Terms: conditions — Brain Neoplasms; Glioma; Glioblastoma; Gliosarcoma | interventions — Erlotinib Hydrochloride; Cytoreduction Surgical Procedures

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- No cytoreductive surgery planned (Experimental): Patients who are not candidates for surgery as part of their routine care will enroll into the medical arm of the trial. They will initiate pulsatile erlotinib dosing and continue therapy until either disease progression or intolerable toxicity.
  Interventions: Drug: erlotinib
- Cytoreductive surgery planned (Experimental): Patients scheduled for "salvage" resection as part of their routine care will be considered for this cohort. They will receive 1 pre-operative dose of 2000 mg erlotinib. Resection will occur ≤ 3 hours after the pre-operative dose. After recovery from surgery, patients will resume pulsatile erlotinib dosing.
  Interventions: Drug: erlotinib; Procedure: Cytoreductive Surgery

INTERVENTIONS:
Drug: erlotinib — For patients with no cytoreductive surgery planned, patients will receive single-agent erlotinib at a starting dose of 2000 mg on days 1 of every 7 days. For patients with cytoreductive surgery planned, patients will receive single-agent erlotinib at a starting dose of 2000 mg day 1 of every 7 days (+/- 2 days). One pre-operative dose of 2000 mg erlotinib will be administered in an open-label, unblinded manner, administered in the hospital "on call" to the operating room.
  Other Names: Tarceva
Procedure: Cytoreductive Surgery — Standard procedure
  Arms: Cytoreductive surgery planned

SUMMARY:
The purpose of this study is to test the effectiveness of a drug called erlotinib in treating the tumor. This is a multi-center pilot study that explores efficacy and molecular effects of high dose weekly erlotinib for recurrent EGFR vIII mutant malignant gliomas, and correlate molecular profile of pre-treatment tissue with outcome.

DETAILED DESCRIPTION:
This is a pilot study of erlotinib for subjects who have a brain tumor called a glioblastoma or another malignant glioma, which has continued to grow after treatment. The purpose of this study is to test the effectiveness of a drug called erlotinib in treating the tumor. The study drug, erlotinib (also called Tarceva) is a pill (taken by mouth) that has been approved by the U.S. Food and Drug Administration (FDA) for the subjects with other cancers (lung cancer or pancreatic cancer). It is not approved for glioblastoma or another malignant glioma. Erlotinib blocks a messenger that tells cancer cells to grow. That messenger is called Epidermal Growth Factor Receptor (EGFR). This type of tumor contains a form of EGFR called variant number 3 (abbreviated EGFR variant III or EGFRvIII for short) that is different from the normal form.Research suggests that erlotinib is particularly effective at stopping EGFRvIII. Research also suggests that high doses of erlotinib taken once per week may be more effective than low doses of erlotinib taken once per day.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed intracranial malignant glioma of the following types: Glioblastoma (GBM), Gliosarcoma (GS), Anaplastic astrocytoma (AA), Anaplastic oligodendroglioma (AO), Anaplastic oligoastrocytoma (AOA, also called anaplastic mixed gliomas or AMG), High grade glioma not otherwise specified (NOS).
* EGFRvIII mutation detected on pretreatment tissue from at least 1 prior surgery.
* At least 15 unstained slides or at least 1 tissue blocks must be collected from at least one prior surgery.
* Recovered from toxic effects of prior therapies.
* Able to undergo contrast enhanced MRI scans (or CT scans for patients unable to tolerate MRI).
* Shown unequivocal evidence for contrast enhancing tumor progression by MRI (or CT for patients who cannot tolerate MRI) in comparison to a prior scan.
* Age > or = 18 years.
* Karnofsky Performance Status > or = 60%.
* Life expectancy of > 8 weeks.
* Normal organ and marrow function, adequate liver function and adequate renal function before starting therapy.
* Women of child-bearing potential and men must agree to use adequate contraception.
* Women of childbearing potential must have a negative pregnancy test documented within 7 days prior to treatment.
* Women must agree not to breast feed.
* Ability to understand and the willingness to sign a written informed consent document.
* Ability to swallow the tablets.

Cohort A (medical) specific inclusion criteria:

* Fulfill all of the general inclusion criteria.
* MRI/CT must demonstrate measurable enhancing tumor of at least 1cm2 in cross-sectional area to allow assessment of radiographic response, unless: measurable disease is not present because the patient underwent gross total resection as the most recent anti-tumor therapy.
* At least 3 months have elapsed between any prior brain radiotherapy and initiation of study therapy.
* MRI/CT must demonstrate measureable enhancing tumor at least 1cm by 1cm squared in cross-sectional area to allow assessment of radiographic response.
* Stable or decreasing dose of corticosteroids for a minimum of 5 days before the baseline MRI/CT.
* The baseline MRI/CT must be performed on the 14th day or less prior to initiation of study treatment.

Cohort B (surgical) specific inclusion criteria:

* Fulfill all of the general inclusion criteria.
* An MRI/CT scan showing progression is required.

Exclusion Criteria:

* Received prior treatment with convection enhanced delivery, other catheter based intratumoral treatment, or carmustine (BCNU)/Gliadel wafers.
* Prior therapy that included stereotactic radiosurgery during therapy for newly diagnosed or recurrent disease, or re-irradiation of any type, must have confirmation of true progressive disease rather than radiation necrosis based upon surgical documentation of recurrent/progressive disease.
* Prior treatment with an EGFR inhibitor.
* Received prior treatment with direct Vascular endothelial growth factor (VEGF)/Vascular Endothelial Growth Factor Receptors (VEGFR) inhibitors.
* Smoking or plan to smoke tobacco or marijuana during study therapy.
* Receiving any other investigational agents concurrently with study treatment.
* Taking Enzyme Inducing Anti-Epileptic Drug (EIAED). If previously on an EIAED, the patient must be off of it for at least two weeks prior to study treatment.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to erlotinib.
* Uncontrolled intercurrent illness that would limit compliance with study requirements.
* Have HIV and are receiving combination antiretroviral therapy.
* Other active concurrent malignancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2011-01-07 (Actual); Primary Completion 2016-11-22 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Clinical Benefit Rate (either radiographic response or at least 6 months of progression-free survival) | Up to 3 years
  All patients will have their tumor measurements recorded at baseline and at the time of each MRI/CT scan.
  Clinical efficacy of pulsatile dosing with the EGFR Tyrosine Kinase Inhibitor erlotinib in patient with EGFR vIII mutant, recurrent malignant gliomas will be explored by determination of radiographic response and 6 month progression-free survival (6mPFS rate).

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Lassman, MD, Principal Investigator — Columbia University
Locations (4):
- United States (4):
  - Memorial Sloan-Kettering at Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan-Kettering Cancer Center at Commack, Commack, New York
  - Columbia University Irving Medical Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm
- See also: AAAJ7500 — http://hiccc.columbia.edu/clinicaltrials/